CLINICAL TRIAL: NCT00438503
Title: Effect of Glucose in Dialysis Water in Diabetics With Chronic Renal Failure on Blood Pressure, Pulse Rate, Plasma Glucose, Plasma Concentrations of Insulin, Growth Hormone, Renin, Angiotensin II, Endothelin and Body Temperature
Brief Title: Glucose in Dialysis Water in Diabetics With Chronic Renal Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MED.RES.2007.02.EBP
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2007-09

CONDITIONS: Renal Failure, Chronic; Diabetic Nephropathies
Keywords: Hemodialysis, diabetes mellitus,; Chronic renal failure, dialysis ,
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetic Nephropathies; Diabetes Mellitus | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Procedure

SUMMARY:
The purposes are 1. to measure the effect of dialysis with glucose in dialysis water on blood pressure, pulse rate, plasma concentration of glucose, plasma concentrations og insulin, glucagon, growth hormone, renin, angiotensin II, endothelin and body temperature, and 2. to analyse the relationship between the changes in blood pressure and changes in vasoactive hormones

DETAILED DESCRIPTION:
The relationship between blood pressure during dialysis treatment and vasoactive hormones are studied. This includes measurements of plasma concentration of glucose, plasma concentrations og insulin, glucagon, growth hormone, renin, angiotensin II, endothelin

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years,
2. Both men and women,
3. Dialysis treatment for at least three month due to diabetic nephropathy

Exclusion Criteria:

1. Heart failure,
2. Lung insufficiency,
3. Chronic liver disease,
4. Malignant disease,
5. Nephrotic syndrome,
6. Lack of compliance,
7. Unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Effect og glucose in dialysis water on blood pressure, plasma glucose and hormones in plasma

SECONDARY OUTCOMES:
Relationship between changes in blood pressure and and changes in hormones

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Regional Hospital Holstebro
Locations (1):
- Holstebro Hospital, Holstebro, Denmark